CLINICAL TRIAL: NCT04127019
Title: Adjuvant Six Cycles of Docetaxel and Cyclophosphamide or Three Cycles of Cyclophosphamide/Epirubicin/Fluorouracil Followed by Three Cycles of Docetaxel Versus Four Cycles of Epirubicin and Cyclophosphamide Followed by Weekly Paclitaxel in Operable Breast Cancer
Brief Title: Adjuvant 6 Cycles of Docetaxel and Cyclophosphamide or 3 Cycles of Cyclophosphamide/Epirubicin/Fluorouracil Followed by 3 Cycles of Docetaxel Versus 4 Cycles of Epirubicin and Cyclophosphamide Followed by Weekly Paclitaxel in Operable Breast Cancer (MASTER)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASTER
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Primary Breast Cancer
MeSH Terms: interventions — Paclitaxel; Docetaxel; Cyclophosphamide; Epirubicin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Experimental: Arm 1 6 cycles of (Docetaxel 75mg/m2 ivgtt d1+ Cyclophosphamide 600 mg/m2 iv d1, 21 days per cycle) .
  Experimental: Arm 2 3 cycles of FEC (Epirubicin 100 mg/m2 ivgtt d1+Cyclophosphamide 500 mg/m2 iv d1+ 5-fluorouracil 500 mg/m2 iv d1, 21 days per cycle) followed by 3 cycles of Docetaxel (Docetaxel 100mg/m2, ivgtt d1, 21 days per cycle)
  Experimental: Arm 3 4 cycles of EC (Epirubicin 90 mg/m2 ivgtt d1+Cyclophosphamide 600 mg/m2 iv d1+ , 21 days per cycle) followed by 4 cycles of Paclitaxel (Paclitaxel 80mg/m2, ivgtt d1,8,15, 21days per cycle).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TC*6 (Experimental): 6 cycles of (Docetaxel 75mg/m2 ivgtt d1+ Cyclophosphamide 600 mg/m2 iv d1, 21 days per cycle) .
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide
- CEF*3-T*3 (Experimental): 3 cycles of CEF (Epirubicin 100 mg/m2 ivgtt d1+Cyclophosphamide 500 mg/m2 iv d1+ 5-fluorouracil 500 mg/m2 iv d1, 21 days per cycle) followed by 3 cycles of Docetaxel (Docetaxel 100mg/m2, ivgtt d1, 21 days per cycle)
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: 5-fluorouracil
- EC*4-wP*12 (Experimental): 4 cycles of EC (Epirubicin 90 mg/m2 ivgtt d1+Cyclophosphamide 600 mg/m2 iv d1, 21 days per cycle) followed by 4 cycles of Paclitaxel (Paclitaxel 80mg/m2, ivgtt d1,8,15, 21days per cycle).
  Interventions: Drug: Paclitaxel; Drug: Cyclophosphamide; Drug: Epirubicin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel chemotherapy (injection)
  Arms: EC*4-wP*12
Drug: Docetaxel — Docetaxel chemotherapy (injection)
  Arms: CEF*3-T*3; TC*6
Drug: Cyclophosphamide — Cyclophosphamide chemotherapy (injection)
Drug: Epirubicin — Epirubicin chemotherapy (injection)
  Arms: CEF*3-T*3; EC*4-wP*12
Drug: 5-fluorouracil — 5-fluorouracil chemotherapy (injection)
  Arms: CEF*3-T*3

SUMMARY:
We aimed to evaluate the noninferiority of a short-term anthracycline-free chemotherapy (TC, six cycles of docetaxel and cyclophosphamide) or a short-term anthracycline-based chemotherapy (CEF-T, three cycles of cyclophosphamide/epirubicin/fluorouracil followed by three cycles of docetaxel) to a standard anthracycline/taxane-containing chemotherapy (EC-P, epirubicin and cyclophosphamide for four cycles followed by paclitaxel for twelve weeks) in operable breast cancer.

DETAILED DESCRIPTION:
It was initiated as an adjuvant chemotherapy trial in 2010 to test noninferiority of an anthracycline-free short-term regimen (T75C600 x 6 [TC] once every 3 weeks) or a short-term regimen (C500E100F500 x 3 once every 3 weeks followed by T100 x 3 every 3 weeks [CEF-T]) compared with a standard long-term anthracycline-containing regimen (E90C600 x 4 once every 3 weeks followed by P80 x 12 once every week [EC-P]). Patients were randomly assigned (1:1:1) to each arm after completing surgical excision of primary tumor. Trastuzumab was administered in combination with chemotherapy to patients with HER2-positive breast cancer and sustained monotherapy as per the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 - 75 years
* Histological confirmed unilateral primary invasive carcinoma of the breast
* Adequate surgical treatment with complete resection of the tumor (R0) and resection of > or = 10 axillary nodes or SLN in clinically N0 patients
* Node positive disease or node negative disease with at least one other risk factor (tumor size > or = 2 cm, grade > or = II)
* No evidence for distant metastasis (M0) after conventional staging
* Performance Status ECOG < or = 1
* The patient must be accessible for treatment and follow-up
* LVEF> 50%
* Negative pregnancy test (urine or serum) within 7 days prior to randomization in premenopausal patients
* Leucocytes > or = 4 x 10^9/L
* platelets > or = 100 x 10^9/L
* haemoglobin > or = 9 g/dL
* total bilirubin < or = 1.5 UNL
* ASAT (SGOT) and ALAT (SGPT) < or = 2.5 UNL
* creatinine < 175 mmol/L (2 mg/dL)

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy）;
2. Has bilateral breast cancer;
3. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
4. Has metastic (Stage 4) breast cancer;
5. Has any >T4 lesion (UICC1987) (with skin involvement, mass adhesion and fixation, and inflammatory breast cancer);
6. Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
7. Patients participating in other clinical trials at the same time;
8. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
9. Has known allergy to taxane and excipients;
10. Has severe or uncontrolled infection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2079 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 5 year

SECONDARY OUTCOMES:
distant disease-free survival | 5 year
overall survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No